CLINICAL TRIAL: NCT04488003
Title: A Two-Part, Phase II, Multi-center Study of the ERK Inhibitor Ulixertinib (BVD-523) for Patients With Advanced Malignancies Harboring MEK or Atypical BRAF Alterations
Brief Title: Study of Ulixertinib for Patients With Advanced Malignancies Harboring MEK or Atypical BRAF Alterations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment challenges
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BVD-523-ABC
Expanded Access: NCT04566393 (Available)
Record Dates: First submitted 2020-07-17; First posted 2020-07-27 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor; BRAF Gene Mutation; BRAF Gene Alteration; MEK Mutation; MEK Alteration; MAP2K1 Gene Mutation; MAP2K1 Gene Alteration; MAP2K2 Gene Mutation; MAP2K2 Gene Alteration
Keywords: atypical BRAF, non-V600
MeSH Terms: interventions — ulixertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Ulixertinib (Experimental): Oral, 600 mg, twice daily, for 28-days in each treatment cycle
  Interventions: Drug: Ulixertinib
- Part B: Ulixertinib (Experimental): Oral, 600 mg, twice daily, for 28-days in each treatment cycle
  Interventions: Drug: Ulixertinib
- Part B: Physician's choice of treatment (Experimental): Physician's choice will be restricted to two approved (not off-label) treatments for each tumor histology (agents targeting BRAF or MEK kinases and experimental agents are not permitted as physician choice). If a patient progresses on physician's choice of treatment, crossover to the ulixertinib arm is permitted.
  Interventions: Drug: Physician's Choice

INTERVENTIONS:
Drug: Ulixertinib — Oral, 600 mg, twice daily, for 28-days in each treatment cycle
  Other Names: BVD-523, BVD523
  Arms: Part A: Ulixertinib; Part B: Ulixertinib
Drug: Physician's Choice — Physician's choice will be restricted to two approved (not off-label) treatments for each tumor histology (agents targeting BRAF or MEK kinases and experimental agents are not permitted as physician choice)).
  Arms: Part B: Physician's choice of treatment

SUMMARY:
This BVD-523-ABC study builds on the safety and clinical activity experience of previous studies that have evaluated ulixertinib as a novel targeted cancer treatment in cohorts of patients with specific genetic alterations and tumor histologies that result in aberrant MAPK pathway signaling. Early clinical data have demonstrated anti-tumor activity with ulixertinib treatment and have identified specific groups of patients for whom additional development is warranted.

DETAILED DESCRIPTION:
This multi-center, phase II study will be conducted in two parts and assess the clinical benefit, safety, pharmacokinetics, and pharmacodynamics of ulixertinib (BVD-523) in patients with advanced malignancies.

Part A (tumor histology agnostic) will be open label and enroll patients to one of six groups based on their tumor alteration. Targeted enrollment per group was 38 patients with a total targeted enrollment of 228 patients. Actual enrollment was total of 104 patients with 77 patients allocated to treatment.

* Group 1: Patients with tumors, other than colorectal cancer (CRC), having a BRAF alteration that results in an amino acid change at positions G469, L485, or L597.
* Group 2: Patients with tumors, other than CRC, having a defined Class 2 BRAF alteration (see Appendix 2 of protocol).
* Group 3: Patients with tumors, other than CRC, having an atypical BRAF alteration (non V600) that is not specified in Group 1 or Group 2.
* Group 4: Patients with CRC having any atypical BRAF alteration.
* Group 5: Patients with tumors, other than CRC, harboring alterations in MEK1/2.
* Group 6: Patients with CRC harboring alterations in MEK1/2.

Part B (tumor histology specific) will randomly enroll patients with one of up to three specified tumor histologies to receive either ulixertinib or the physician's choice of treatment in a 2:1 ratio. Tumors must harbor a specified MEK or atypical BRAF alteration. If a patient progresses on physician's choice of treatment, crossover to the ulixertinib arm is permitted.The specific histologies to be included in this part will be selected based on available data and discussion with the clinical investigators, the medical monitor, and the sponsor. Total enrollment was targeted to approximately 80-100 patients per histology with up to three histologies included; however, the study was terminated prior to any patients enrolling in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a locally advanced or metastatic malignancy, that has progressed following systemic therapy for their disease, if available, or for which the patient is not a candidate or refuses.
* Tumors harboring a MEK or atypical BRAF alteration.
* Provide signed and dated informed consent prior to initiation of any study-related procedures that are not considered standard of care (SoC).
* Male or female patients aged ≥18 years.
* Patients must have measurable disease by RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
* Adequate renal function [creatinine ≤1.5 times ULN (upper limit of normal)] or a glomerular filtration rate (GFR) of ≥50 mL/min (using Cockcroft-Gault).
* Adequate hepatic function [total bilirubin ≤1.5 times ULN; AST (aspartate transaminase) and ALT (alanine transaminase) ≤3 times ULN or ≤5 times ULN if the elevation is due to liver involvement by tumor].
* Adequate bone marrow function (hemoglobin ≥9.0 g/dL; platelets ≥100 x 109 cells/L; absolute neutrophil count ≥1.5 x 109 cells/L).
* Adequate cardiac function: Left ventricular ejection fraction (LVEF) of >50% as assessed by multi-gated acquisition (MUGA) or ultrasound/echocardiography (ECHO); and a corrected QT interval (QTc) <480ms by the Fridericia method (QTcF).
* Contraception - women: Negative pregnancy test for females of child-bearing potential; must be surgically sterile, postmenopausal (no menstrual cycle for at least 12 consecutive months), or compliant with a medically approved contraceptive regimen during and for 3 months after the last administration of study drug. Abstinence is not considered an adequate contraceptive regimen.
* Contraception - men: Must be surgically sterile, or compliant with a medically approved contraceptive regimen during and for 3 months after the last administration of study drug.
* Willing and able to participate in the trial and comply with all trial requirements.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational agent may be included after consultation with the medical monitor.

Exclusion Criteria:

* Gastrointestinal (GI) condition that could impair absorption of study medication (specific cases e.g., remote history of GI surgery, may be enrolled after discussion with the medical monitor) or inability to ingest study medication.
* Uncontrolled or severe intercurrent medical condition.
* Known uncontrolled brain metastases. Stable brain metastases either treated or being treated with a stable dose of steroids/anticonvulsants, with no dose change in the previous 4 weeks, can be allowed.
* Having received any cancer-directed therapy (chemotherapy, hormonal therapy, biologic or immunotherapy, etc.) within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. Patients previously treated with radiotherapy must have recovered from the acute toxicities associated with such treatment.
* Major surgery within 4 weeks prior to first dose.
* Any use of an investigational drug within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. A minimum of 10 days between termination of the prior investigational drug and administration of study drug is required. In addition, any drug-related toxicity except alopecia should have recovered to Grade 1 or less.
* Prior therapy with any ERK inhibitor (e.g. LY3214996, LTT462).
* Groups 1-4: Prior therapy with any BRAF and/or MEK inhibitor (e.g. encorafenib, dabrafenib, vemurafenib, binimetinib, trametinib, cobimetinib) is excluded. Prior BRAF and/or MEK inhibitor therapy is permitted for Groups 5 and 6.
* For Part B, agents targeting BRAF or MEK kinases and experimental agents are not permitted as physician's choice
* Pregnant or breast-feeding women.
* Any evidence of serious active infections. Patients are allowed to enroll if they have been fever-free for at least 48 hours and are on an active treatment that is not prohibited in Appendix 1 of the protocol.
* Any important medical illness or abnormal laboratory finding that would increase the risk of participating in this study (based on the investigator's judgment).
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* Concurrent therapy with any other investigational agent.
* Concurrent therapy with drugs known to be strong inhibitors or inducers of CYP1A2, CYP2D6, and CYP3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Mayo Clinic, Phoenix, Arizona
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Christiana Care Health Services / Helen F. Graham Cancer Center, Newark, Delaware
  - Johns Hopkins Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota Community Oncology Research Consortium (MMCORC), Saint Louis Park, Minnesota
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center / Duke Cancer Institute, Durham, North Carolina
  - Kettering Cancer Center, Kettering, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC - Sarah Cannon (SCRI), Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Germann UA, Furey BF, Markland W, Hoover RR, Aronov AM, Roix JJ, Hale M, Boucher DM, Sorrell DA, Martinez-Botella G, Fitzgibbon M, Shapiro P, Wick MJ, Samadani R, Meshaw K, Groover A, DeCrescenzo G, Namchuk M, Emery CM, Saha S, Welsch DJ. Targeting the MAPK Signaling Pathway in Cancer: Promising Preclinical Activity with the Novel Selective ERK1/2 Inhibitor BVD-523 (Ulixertinib). Mol Cancer Ther. 2017 Nov;16(11):2351-2363. doi: 10.1158/1535-7163.MCT-17-0456. Epub 2017 Sep 22. PMID 28939558
- [Background] Sullivan RJ, Infante JR, Janku F, Wong DJL, Sosman JA, Keedy V, Patel MR, Shapiro GI, Mier JW, Tolcher AW, Wang-Gillam A, Sznol M, Flaherty K, Buchbinder E, Carvajal RD, Varghese AM, Lacouture ME, Ribas A, Patel SP, DeCrescenzo GA, Emery CM, Groover AL, Saha S, Varterasian M, Welsch DJ, Hyman DM, Li BT. First-in-Class ERK1/2 Inhibitor Ulixertinib (BVD-523) in Patients with MAPK Mutant Advanced Solid Tumors: Results of a Phase I Dose-Escalation and Expansion Study. Cancer Discov. 2018 Feb;8(2):184-195. doi: 10.1158/2159-8290.CD-17-1119. Epub 2017 Dec 15. PMID 29247021
- See also: BioMed Valley Discoveries — https://biomed-valley.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 24 clinical sites in the USA. Enrollment took place between January 2021 and December 2022.
Period: Assessed for Eligibility
Arm/Group | Part A: Ulixertinib | Part B: Ulixertinib | Part B: Physician's Choice of Treatment
Started | 104 | 0 | 0
Completed | 77 | 0 | 0
Not Completed | 27 | 0 | 0
Not completed — Screen Failure | 24 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Allocated to Treatment
Arm/Group | Part A: Ulixertinib | Part B: Ulixertinib | Part B: Physician's Choice of Treatment
Started | 77 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 77 | 0 | 0
Not completed — Progressive Disease | 51 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Other | 5 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0
Not completed — Death | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Part A: Ulixertinib
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 70
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 77
ECOG Performance at Baseline [Count of Participants; unit: Participants] — ECOG performance status was assessed by the clinical site investigator/physician or their designee; ECOG 0 - Fully active, able to carry on all pre-disease performance without restriction; ECOG 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; ECOG 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  Participants
    ECOG 0 | 23
    ECOG 1 | 50
    ECOG 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part A: Overall Response Rate (ORR) According to RECIST 1.1
Description: ORR will be defined as the percentage of patients achieving a Best Overall Response (BOR) of confirmed Complete Response (CR) and/or Partial Response (PR). Patients will be evaluated at baseline & at periodic follow-up visits through the time their participation in the study is complete.The best responses will occur at different time points for each patient.
Time Frame: Up to 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Ulixertinib
Number analyzed (Participants) | 77
Participants | 0

2. Secondary Outcome: Part A: Progression Free Survival (PFS) According to RECIST 1.1
Description: PFS will be defined as time from first day of study drug to disease progression or death. Patients with no event will be censored at the last available tumor assessment. This analysis will be based on investigator assessment.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: Ulixertinib
Number analyzed (Participants) | 66
months | 1.5 [1.0 to 2.5]

3. Secondary Outcome: Part A: Overall Survival (OS) According to RECIST 1.1
Description: OS will be defined as time from first day of study drug to death. Patients with no event will be censored at the last date the patient is known to be alive.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: Ulixertinib
Number analyzed (Participants) | 50
months | 5.2 [3.8 to 7.0]

4. Secondary Outcome: Part A: Pharmacokinetic Concentration of BVD-523 at Steady State
Description: Single time point taken prior to taking study drug (trough) at steady state. Steady state is defined as patients who have received at least 5 days, or 10 consecutive doses, of study drug.
Time Frame: Single time point drawn at Visit 4/approximately day 15 (or whenever the patient reaches steady state).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Ulixertinib
Number analyzed (Participants) | 40
ng/mL | 1136.39 (689.538)

ADVERSE EVENTS:
Time Frame: All reportable events were recorded with start dates occurring any time after informed consent obtained through and including 30 calendar days after the last administration of ulixertinib, an average of 2.72 months per patient. If the patient begins a new anti-cancer therapy, the safety reporting period ends at the time the new treatment is started, however, death must always be reported when it occurs during the 30-day reporting period irrespective of intervening treatment.
Description: If there is more than one medical history within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one medical history within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.
  AEs were collected/assessed at each study visit.
Arm/Group | Part A: Ulixertinib
All-Cause Mortality (participants affected / at risk) | 52/104
Serious Adverse Events (participants affected / at risk) | 41/77
Other Adverse Events (participants affected / at risk) | 76/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Ulixertinib (N=77)
Disease progression (General disorders) | 14
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Anorectal infection bacterial (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 2
Cauda equina syndrome (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Postrenal failure (Renal and urinary disorders) | 1
Gallbladder rupture (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mental status changes (Psychiatric disorders) | 2
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Ulixertinib (N=77)
Diarrhoea (Gastrointestinal disorders) | 35
Nausea (Gastrointestinal disorders) | 35
Vomiting (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 28
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 5
Fatigue (General disorders) | 23
Oedema peripheral (General disorders) | 16
Disease progression (General disorders) | 14
Pyrexia (General disorders) | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20
Decreased appetite (Metabolism and nutrition disorders) | 17
Hyponatraemia (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Blood creatinine increased (Investigations) | 20
Aspartate aminotransferase increased (Investigations) | 12
Alanine aminotransferase increased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 4
Weight decreased (Investigations) | 4
Anaemia (Blood and lymphatic system disorders) | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Urinary tract infection (Infections and infestations) | 12
Pneumonia (Infections and infestations) | 6
Rash pustular (Infections and infestations) | 4
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 6
Syncope (Nervous system disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 4
Haematuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 4
Vision blurred (Eye disorders) | 4
Insomnia (Psychiatric disorders) | 6
Hypotension (Vascular disorders) | 8
Hypertension (Vascular disorders) | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Tachycardia (Cardiac disorders) | 6

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of patients analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04488003/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT04488003/SAP_001.pdf